CLINICAL TRIAL: NCT01712256
Title: Re-boosting of Subjects Previously Included in the CT BI-Vacc-4x 2007/1 Study. An Open, Multicenter, Immunogenicity, Follow-up Re-boosting Study With Vacc-4x in Subjects Infected With HIV-1 Who Have Maintained an Adequate Response to ART
Brief Title: Re-boosting of HIV-1 Infected Subjects With Vacc-4x
Acronym: Re-boost
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bionor Immuno AS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-BI Vacc-4x 2012/1
Record Dates: First submitted 2012-10-16; First posted 2012-10-23 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: HIV-1 Infection
Keywords: CD4; Clinical trial; Human immunodeficiency virus-1 (HIV-1); HIV; Immunomodulary; Infection; Phase II; Re-boost; Vaccine; Vacc-4x
MeSH Terms: conditions — Infections | interventions — Vacc-4x

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Re-boosting with Vacc-4x (Experimental): Intradermal Vacc-4x (1.2 mg) given with Leukine® (rhu-GM-CSF) (0.06 mg) at day 1 and day 15.
  Interventions: Biological: Vacc-4x

INTERVENTIONS:
Biological: Vacc-4x — Vacc-4x is a peptide-based HIV immunotherapy administered intradermally. Vacc-4x peptides are reconstituted in sterile water.
  Other Names: Combination of Vacc-10, Vacc-11, Vacc-12 and Vacc-13

SUMMARY:
During the course of HIV infection the number of CD4 cells decreases, resulting in a reduced immunological response and eventually immune deficiency. Vacc-4x is a peptide-based HIV immunotherapy vaccine and is anticipated to strengthen the immune system's response to HIV.

All patients participating in this trial have previously received the vacc-4x vaccine in order to reduce the amount of HIV-1 virus in the blood and increase the immune response. The primary objective of this study is to evaluate if a re-boost with Vacc-4x could further reduce the amount of HIV-1 virus and increase the immune response.

DETAILED DESCRIPTION:
Human immunodeficiency virus (HIV) infects the cluster of differentiation 4 (CD4) subset of T-cells that are critical for initiating immune responses to infection. The level of CD4 cells in the blood is a marker of a patient's immunological status. During the course of an HIV infection, the number of CD4 cells decreases, resulting in reduced immunological responsiveness and ultimately immune deficiency.

Current management of an HIV infection includes antiretroviral therapy (ART). The advent of effective ART in 1996 led to a profound decrease in type 1 HIV (HIV-1)-associated morbidity and mortality in developed countries where ART has been available.

Despite the ability of ART to inhibit HIV-1 replication, it cannot cure infection, making ART a lifelong treatment that requires sustained compliance and imposes significant individual and societal financial burdens on healthcare services. Furthermore, ART side effects (e.g., metabolic toxicity and stigmatizing body fat redistribution) often require medication that further increases the inconveniences and financial burdens of HIV management. Of additional concern is the emergence of viruses resistant to ART that can result in treatment failure.

Vacc-4x is a peptide-based HIV therapeutic vaccine. The primary objective of Vacc-4x therapeutic vaccine is to strengthen the immune system's response to HIV p24. ART dramatically reduces the level of virus in circulation in the body, thereby allowing the immune system to focus on the therapeutic vaccine that is administered. ART also allows for the generation of new naïve CD4 cells that can be triggered by the therapeutic vaccine to generate new immune responses to HIV-1. Subjects are therefore immunized with Vacc-4x in the presence of ART to generate new HIV-specific immune responses that can sustain immunological fitness for prolonged periods when patients are removed from ART. It is likely that periodic boosting on ART will be required to sustain the immunotherapeutic effect - in this way ART may become an intermittent therapy.

This study is a follow-up, re-boosting study of Study CT-BI Vacc-4x 2007/1 (EudraCT Number 2007-006302-13) performed in US and Europe (UK, Germany, Spain and Italy). All subjects to be included have been given a therapeutic immunization with Vacc-4x during the CT-BI Vacc-4x 2007/1 study. During the study a reduction in the viral load set-point (mean viral load at Week 48 and Week 52, or if Week 52 not reached, mean viral load of the last two measured values before restart of ART) was seen in the Vacc-4x group compared to placebo group. Further stimulation of the immune system by re-boosting with Vacc-4x could reduce the viral load set-point further.

ELIGIBILITY:
Inclusion Criteria:

1. Completed immunization regimen with Vacc-4x active and stopped ART (at Week 28) in the CT-BI Vacc-4x 2007/1 study. (No re-start of ART is required).
2. Documented pre-study CD4 cell count ≥400x106/L.
3. Documented pre-study viral load < 300 000copies/mL.
4. Signed informed consent.

Exclusion Criteria:

1. Reported AIDS-defining illness within the previous year.
2. Malignant disease.
3. On chronic treatment with immune-suppressive therapy.
4. Unacceptable values of the hematologic and clinical chemistry parameters, as judged by the Investigator, including creatinine values >1.5 x upper limit of normal (ULN), and AST, ALT and alkaline phosphatase (ALP) values >2.5 x ULN.
5. Concurrent chronic active infection such as viral hepatitis B or C or tuberculosis.
6. Pregnant or breastfeeding women.
7. Women of childbearing potential not using reliable and adequate contraceptive methods (defined as: use of oral, implanted, injectable, mechanical or barrier products for the prevention of pregnancy; practicing abstinence; sterile) during the 5 weeks re-boosting period including the DTH and for 2 weeks after the DTH test, or sexually active male subjects with partners of child bearing potential unwilling to practice effective contraception during the 5 weeks re-boosting period including the DTH and for 12 weeks after the DTH-test.
8. Current participation in other clinical therapeutic studies.
9. Incapability of compliance to treatment protocol, in the opinion of the Investigator.

Ages: 18 Years to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2012-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vidar Wendel-Hansen, Dr. med, Study Director — Bionor Pharma ASA, Kronprinsesse Märthas Plass 1, P.O. Box 1477 Vika, NO-0116 Oslo, Norway
Locations (10):
- United States (2):
  - UCLA CARE Center, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
- Germany (4):
  - Universitätsklinikum Bonn, Medizinische Klinik und Poliklinik I; Immunologische Ambulanz, Siegmund-Freud-Str. 25, Bonn, Bonn
  - ifi - Studien und Projekte GmbH, an der Asklepios-Klinik St. George, Hamburg, Hamburg
  - EIPMED - Gesellschaft fűr epidemiologische und klinische Forschung in der Medizin mbH Rubensstrasse 125, Berlin, State of Berlin
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
- Istituto San Raffaele, Milan, Milano, Italy
- Spain (2):
  - Hospital Germans Trias i Pujol, Badalona
  - Unidad de VIH, Hospital de Bellvitge, Calle Feixa Llarga s/n, Hospitalet de Llobregat., Barcelona
- Harrison Wing St Thomas' Hospital, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Participants have not provided informed consent for their anonymized individual data to be made available beyond that described in the patient information sheet.

REFERENCES:
- [Background] Kran AM, Sommerfelt MA, Baksaas I, Sorensen B, Kvale D. Delayed-type hypersensitivity responses to HIV Gag p24 relate to clinical outcome after peptide-based therapeutic immunization for chronic HIV infection. APMIS. 2012 Mar;120(3):204-9. doi: 10.1111/j.1600-0463.2011.02843.x. Epub 2011 Nov 27. PMID 22339677
- [Background] Lind A, Sommerfelt M, Holmberg JO, Baksaas I, Sorensen B, Kvale D. Intradermal vaccination of HIV-infected patients with short HIV Gag p24-like peptides induces CD4 + and CD8 + T cell responses lasting more than seven years. Scand J Infect Dis. 2012 Aug;44(8):566-72. doi: 10.3109/00365548.2011.653581. Epub 2012 Feb 19. PMID 22339485
- [Background] Jones T. Vacc-4x, a therapeutic vaccine comprised of four engineered peptides for the potential treatment of HIV infection. Curr Opin Investig Drugs. 2010 Aug;11(8):964-70. PMID 20721838
- [Background] Kran AM, Sorensen B, Sommerfelt MA, Nyhus J, Baksaas I, Kvale D. Long-term HIV-specific responses and delayed resumption of antiretroviral therapy after peptide immunization targeting dendritic cells. AIDS. 2006 Feb 28;20(4):627-30. doi: 10.1097/01.aids.0000210620.75707.ac. PMID 16470131
- [Derived] Rockstroh JK, Asmuth D, Pantaleo G, Clotet B, Podzamczer D, van Lunzen J, Arasteh K, Mitsuyasu R, Peters B, Silvia N, Jolliffe D, Okvist M, Krogsgaard K, Sommerfelt MA. Re-boost immunizations with the peptide-based therapeutic HIV vaccine, Vacc-4x, restores geometric mean viral load set-point during treatment interruption. PLoS One. 2019 Jan 30;14(1):e0210965. doi: 10.1371/journal.pone.0210965. eCollection 2019. PMID 30699178

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Re-boosting With Vacc-4x
Started | 33
Completed | 32
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Re-boosting With Vacc-4x
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.0 (7.12)
Gender [Count of Participants; unit: Participants]
  Female | 6
  Male | 27
Region of Enrollment [Number; unit: participants]
  United States | 8
  United Kingdom | 3
  Italy | 2
  Germany | 10
  Spain | 10
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.64 (5.077)
Time since HIV diagnosis [Mean (Standard Deviation); unit: Days] | 5786.8 (2043.44)
Total time on ART [Mean (Standard Deviation); unit: months] | 138.6 (57.42)
Currently on ART [Number; unit: participants] | 30
Pre-ART HIV-1 viral load [Mean (Standard Deviation); unit: copies/mL] — Population: Examination of the data suggest that the CRF question was interpreted in different ways with respect to stopping and starting ART, and changing the composition of the ART received and the answers given cannot be relied upon.
  copies/mL
    number analyzed (Participants) | 27
    (all) | 67502.4 (150008.65)

OUTCOME MEASURES:

1. Primary Outcome: Vacc-4x Effect on Viral Load Set-point
Description: Viral load (VL) set point in the present re-boost study was compared with VL set point in the 2007/1 study.
Time Frame: 37 weeks
Population: In the ITT population there were 20 evaluable subjects out of 30 (3 subjects did not receive ART from Screening through Week 12) and in the PP population there were 18 evaluable subjects out of 27 (an additional 3 subjects did not discontinue ART at Week 12).
Measure: Mean (Standard Deviation); unit: Copies/mL
Arm/Group | Re-boosting With Vacc-4x
Number analyzed (Participants) | 30
Copies/mL
  CT Vacc-4x 2012/1 VL set point, ITT: number analyzed (Participants) | 20
  CT Vacc-4x 2012/1 VL set point, ITT | 38455.0 (46628.69)
  CT Vacc-4x 2012/1 VL set point, PP: number analyzed (Participants) | 18
  CT Vacc-4x 2012/1 VL set point, PP | 40088.8 (48923.00)
  CT-BI Vacc-4x 2007/1 VL Set Point, ITT: number analyzed (Participants) | 22
  CT-BI Vacc-4x 2007/1 VL Set Point, ITT | 45253.9 (55676.68)
  CT-BI Vacc-4x 2007/1 VL Set Point, PP: number analyzed (Participants) | 20
  CT-BI Vacc-4x 2007/1 VL Set Point, PP | 47336.8 (58031.65)

2. Secondary Outcome: Vacc-4x Effect on Immune Response Measured as CD4 Count
Description: Effect of Re-boost with Vacc-4x on immune response obtained following immunization with Vacc-4x in Study CT-BI Vacc-4x 2007/1
Time Frame: 36 weeks
Population: The ITT includes 30 subjects (3 did not receive ART from Scr. through Week 12) and the PP includes 27 (an additional 3 did not discontinue ART at Week 12).
  Due to the influence of ART on efficacy endpoints, certain subjects or part of their data were excluded from the full ITT and PP, based on when they were on or off ART during the study.
Measure: Mean (Standard Deviation); unit: cells/micro liter
Arm/Group | Re-boosting With Vacc-4x
Number analyzed (Participants) | 30
cells/micro liter
  Baseline; ITT: number analyzed (Participants) | 29
  Baseline; ITT | 782.21 (278.303)
  Baseline, PP: number analyzed (Participants) | 27
  Baseline, PP | 795.74 (283.990)
  Week 2, ITT: number analyzed (Participants) | 29
  Week 2, ITT | 764.8 (245.79)
  Week 2, PP: number analyzed (Participants) | 27
  Week 2, PP | 778.1 (731.0)
  Week 4, ITT: number analyzed (Participants) | 29
  Week 4, ITT | 791.1 (321.53)
  Week 4, PP: number analyzed (Participants) | 27
  Week 4, PP | 805.6 (328.31)
  Week 12, ITT: number analyzed (Participants) | 29
  Week 12, ITT | 772.2 (324.2)
  Week 12, PP: number analyzed (Participants) | 27
  Week 12, PP | 789.4 (326.96)
  Week 16, ITT: number analyzed (Participants) | 27
  Week 16, ITT | 705.2 (233.36)
  Week 16, PP: number analyzed (Participants) | 25
  Week 16, PP | 718.1 (235.41)
  Week 20, ITT: number analyzed (Participants) | 27
  Week 20, ITT | 574.9 (185.81)
  Week 20, PP: number analyzed (Participants) | 25
  Week 20, PP | 581.2 (191.63)
  Week 24, ITT: number analyzed (Participants) | 23
  Week 24, ITT | 544.0 (144.60)
  Week 24, PP: number analyzed (Participants) | 21
  Week 24, PP | 557.9 (142.98)
  Week 28, ITT: number analyzed (Participants) | 20
  Week 28, ITT | 534.2 (140.16)
  Week 28, PP: number analyzed (Participants) | 18
  Week 28, PP | 542.5 (145.70)
  Week 36, ITT: number analyzed (Participants) | 3
  Week 36, ITT | 579.0 (59.57)
  Week 36, PP: number analyzed (Participants) | 3
  Week 36, PP | 579.0 (59.57)

3. Secondary Outcome: Vacc-4x Effect on Immune Response Measured as CD8 Count
Description: as for outcome 2
Time Frame: 36 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cells/micro liter
Arm/Group | Re-boosting With Vacc-4x
Number analyzed (Participants) | 30
cells/micro liter
  Baseline; ITT: number analyzed (Participants) | 29
  Baseline; ITT | 979.43 (352.891)
  Baseline, PP: number analyzed (Participants) | 27
  Baseline, PP | 972.19 (364.810)
  Week 2, ITT: number analyzed (Participants) | 29
  Week 2, ITT | 988.7 (315.63)
  Week 2, PP: number analyzed (Participants) | 27
  Week 2, PP | 971.4 (320.59)
  Week 4, ITT: number analyzed (Participants) | 29
  Week 4, ITT | 926.3 (361.44)
  Week 4, PP: number analyzed (Participants) | 27
  Week 4, PP | 919.0 (369.43)
  Week 12, ITT: number analyzed (Participants) | 29
  Week 12, ITT | 952.0 (451.76)
  Week 12, PP: number analyzed (Participants) | 27
  Week 12, PP | 954.0 (455.80)
  Week 16, ITT: number analyzed (Participants) | 27
  Week 16, ITT | 962.6 (307.56)
  Week 16, PP: number analyzed (Participants) | 25
  Week 16, PP | 966.9 (311.06)
  Week 20, ITT: number analyzed (Participants) | 27
  Week 20, ITT | 1282.1 (633.71)
  Week 20, PP: number analyzed (Participants) | 25
  Week 20, PP | 1257.8 (649.42)
  Week 24, ITT: number analyzed (Participants) | 23
  Week 24, ITT | 1430.9 (588.85)
  Week 24, PP: number analyzed (Participants) | 21
  Week 24, PP | 1444.6 (609.71)
  Week 28, ITT: number analyzed (Participants) | 20
  Week 28, ITT | 1261.9 (511.76)
  Week 28, PP: number analyzed (Participants) | 18
  Week 28, PP | 1245.1 (536.84)
  Week 36, ITT: number analyzed (Participants) | 3
  Week 36, ITT | 1230.7 (192.25)
  Week 36, PP: number analyzed (Participants) | 3
  Week 36, PP | 1302.7 (192.25)

4. Secondary Outcome: Delayed Type Hypersensitivity Test (DTH), Positive Responses for Induration
Description: The proportion of subjects who show Delayed Type Hypersensitivity (DTH) during the treatment phase.
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Re-boosting With Vacc-4x
Number analyzed (Participants) | 30
participants
  Week 0, ITT | 10
  Week 0, PP: number analyzed (Participants) | 27
  Week 0, PP | 9
  Week 4, ITT | 20
  Week 4, PP: number analyzed (Participants) | 27
  Week 4, PP | 19

5. Secondary Outcome: Delayed Type Hypersensitivity Test (DTH), Positive Responses for Erythema
Description: The proportion of subjects who show Delayed Type Hypersensitivity (DTH) during the treatment phase.
Time Frame: 4 Weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Re-boosting With Vacc-4x
Number analyzed (Participants) | 30
participants
  Week 0, ITT | 19
  Week 0, PP: number analyzed (Participants) | 27
  Week 0, PP | 17
  Week 4, ITT | 19
  Week 4, PP: number analyzed (Participants) | 27
  Week 4, PP | 18

6. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: To evaluate the safety and tolerability of re-boosting with Vacc-4x by number of participants with Adverse Events
Time Frame: 37 weeks
Measure: Number; unit: participants
Arm/Group | Re-boosting With Vacc-4x
Number analyzed (Participants) | 33
participants
  With any TEAE | 31
  With injection site reaction | 19
  With any TESAE | 2
  With any AE leading to discontinuation | 0
  Deaths | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of written informed consent until completion of the study at Visit 10.
Arm/Group | Re-boosting With Vacc-4x
Serious Adverse Events (participants affected / at risk) | 2/33
Other Adverse Events (participants affected / at risk) | 31/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Re-boosting With Vacc-4x (N=33)
HIV infection (Infections and infestations) | 1 (1)
Oropharyngeal cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Re-boosting With Vacc-4x (N=33)
Application site pruritus (General disorders) | 16 (21)
Injection site pruritus (General disorders) | 13 (17)
Fatigue (General disorders) | 7 (8)
Influenza-like illness (General disorders) | 4 (4)
Injection site erythema (General disorders) | 4 (6)
Asthenia (General disorders) | 3 (4)
Application site reaction (General disorders) | 2 (5)
Injection site Vesicles (General disorders) | 2 (3)
Oral candidiasis (Infections and infestations) | 4 (4)
Bronchitis (Infections and infestations) | 2 (2)
Gastroenteritis (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Pain in extremities (Musculoskeletal and connective tissue disorders) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Headache (Nervous system disorders) | 6 (6)
Paraesthesia (Nervous system disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4)
Night sweats (Skin and subcutaneous tissue disorders) | 3 (5)
Lymphadenopathy (Blood and lymphatic system disorders) | 6 (10)
diarrhoea (Gastrointestinal disorders) | 3 (4)
Nausea (Gastrointestinal disorders) | 3 (3)
Aphthous stomatitis (Gastrointestinal disorders) | 2 (3)
Contusion (Injury, poisoning and procedural complications) | 2 (3)
Hypertension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor (or designee) will prepare a final report on the study. The Investigator may not publish or present any information on this study without the express written approval of the Sponsor. Additionally, the Sponsor, may, for any reason, withhold approval for publication or presentation.